CLINICAL TRIAL: NCT06938685
Title: Evaluation of the Efficacy of NeoThelium FT in the Healing of Chronic Diabetic Foot Ulcers: A Randomized Controlled Multicenter Crossover Trial
Brief Title: Evaluating the Efficacy NeoThelium FT in the Treatment of Diabetic Foot Ulcers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NuScience Medical Biologics, LLC (Industry)
Collaborators: SygNola, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OMNEO
Record Dates: First submitted 2025-03-31; First posted 2025-04-22 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Foot Ulcer
Keywords: Chronic wounds; Wound Medicine; Cellular, Acellular, Matrix-like Product (CAMP); Cellular and/or Tissue Product (CTP); Dehydrated Complete Human Placental Membrane (dCHPM)
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The subject will be randomized to one of the following treatments:
  * Standard of care
  * NeoThelium FT in addition to standard of care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention: Standard of Care (Active Comparator): Wound cleansing, Sharps debridement, Dressing for moisture balance, Offloading
  Interventions: Other: Standard of Care
- Intervention: NeoThelium FT & Standard of Care (Experimental): Wound cleansing, sharps debridement, NeoThelium FT application, Dressing for moisture balance, Offloading
  Interventions: Other: NeoThelium FT

INTERVENTIONS:
Other: Standard of Care — Wound cleansing, Sharps debridement, Dressing for moisture balance, Offloading
  Arms: No Intervention: Standard of Care
Other: NeoThelium FT — NeoThelium FT is a dehydrated wound covering derived from donated human placental tissue. NeoThelium FT is a dual-layer membrane with amnion and chorion combination layers.
  Arms: Intervention: NeoThelium FT & Standard of Care

SUMMARY:
This is a randomized controlled crossover trial evaluating the efficacy of NeoThelium FT in conjunction with standard of care vs. standard of care alone in treating diabetic foot ulcers.

DETAILED DESCRIPTION:
This research will take place across multiple medical centers, where both researchers and participants will know which treatment is being used (open label). Patients who agree to participate and meet the study requirements during screening will be randomly assigned to one of two groups: either standard of care (SOC) alone, or SOC plus NeoThelium FT.

The study includes a crossover component for subjects in the SOC arm. At treatment visit 13 (approximately 84 days post-randomization), SOC arm subjects not having achieved complete wound closure, and still meeting the inclusion/exclusion criteria, are eligible to cross over to the IP arm (SOC plus NeoThelium FT). Crossover subjects will begin IP arm treatment with weekly NeoThelium FT applications for up to 12 treatment visits. The subject will continue follow-up per the original schedule. As this is a post-marketing study, it will gather information regarding the efficacy of treatment while also supporting insurance reimbursement decisions. All subjects will complete a two-week screening phase prior to being randomized into a treatment arm. Treatment arms will consist of NeoThelium FT in conjunction with standard of care, vs. standard of care alone. The primary endpoint will be the percentage of target ulcers that achieve complete wound closure within 12 weeks. Secondary endpoints consist of wound area reduction rates, time to closure, follow-up closure, and pain assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, 18 years of age or older
2. Subject has a medical diagnosis of Type I or Type II Diabetes Mellitus requiring oral or glycemic control and/or insulin replacement therapy
3. Subject has a diabetic foot ulcer present for 4 weeks or greater (documented in medical record), and less than 12 months duration if being treated with continuous SOC
4. Subject has a diabetic foot ulcer with a historical wound measurement showing less than 25% healing in 14 days prior to screening
5. Subject has a diabetic foot ulcer with screening wound measurement showing less than 25% healing in 14 days prior to randomization
6. Subject has a diabetic foot ulcer of Wagner grade 1, 2, or 3 without infection or clinically visible exposed bone. Wagner 3 is acceptable if the diagnosis is acute osteomyelitis and the subject has successfully completed IV antibiotic treatment prior to screening.
7. Index ulcer is a minimum of 0.5cm2 and a maximum of 25cm2 at first treatment visit
8. Diabetic foot ulcer is being treated with offloading therapy for 14 days prior to randomization
9. Adequate circulation of ulcer demonstrated by an ABI of >0.7 and <1.3, or TBI of >0.6 within 30 days prior to randomization OR an arterial ultrasound noted with patent circulation and without significant stenosis 90 days prior to randomization.
10. Index ulcer is free of infection prior to randomization and during screening phase. Infection must be adequately treated and controlled as defined by Infectious Disease Society of America (IDSA) Guidelines PEDIS Grade 1.
11. Index ulcer is free of necrotic debris prior to NeoThelium FT application
12. Female subjects of childbearing potential having a negative pregnancy test prior to randomization
13. Subject is able and willing to follow the protocol requirements
14. Subject had signed informed consent
15. If 2 or more ulcers are present, the ulcers must be separated by at least 2 cm

Exclusion Criteria:

1. Subject has a known life expectance of <1 year
2. Subject is unable to comply with protocol treatment
3. Subject has major uncontrolled medical disorders in the opinion of the investigator, such as serious cardiovascular, renal, liver, pulmonary, autoimmune, palliative care, or inherited blood disorders that may affect wound healing
4. Subject actively being treated for malignant disease or history of malignancy or radiation therapy at the site of wound
5. Subject has comorbid conditions that may compromise subject safety in the opinion of the investigator
6. Known contraindications to tissue-engineered allograft
7. Concurrent participation in alternative clinical trial that involves investigational drug or device interfering with wound treatment and/or healing
8. Subject is pregnant or breastfeeding
9. Subject with history of immunosuppressant treatment (systemic corticosteroids >10mg daily dose), cytotoxic chemotherapy, or topical steroid application to the ulcer surface for >2 weeks duration within 30 days prior to randomization; or anticipated use of the above during the course of the study
10. Wound previously treated with CAMPs, tissue engineered, or scaffold materials within 30 days prior to randomization
11. Diabetic foot ulcer of Wagner 3 grade with active acute infection that has not completed IV antibiotic treatment, or Wagner 3 grade with chronic refractory osteomyelitis
12. Wound depth with visible exposed bone
13. HBOT within 14 days prior to randomization
14. Revascularization surgery on the index ulcer leg within 30 days of screening phase
15. Index ulcer suspicious of neoplasm in the opinion of the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Complete Wound Closure | 1-12 weeks
  The primary endpoint will be the percentage of target ulcers that achieve complete wound closure.

SECONDARY OUTCOMES:
Percentage Wound Area Change | 1-12 weeks
  The percentage change in wound area from TV-1 to TV-13 will be measured weekly using digital photographic planimetry and physical examination.
Pain Assessment | Day 0, Day 14, Day 35, Day 56, Day 84
  Change in pain associated with the target ulcer will be assessed using the Numeric Pain Rating Scale at designated time points

OTHER OUTCOMES:
Hemoglobin A1c | Day -14 through 91 days
  Incidence of wound closure vs HbA1c
Adverse Events and Serious Adverse Events | Day -14 through 91 days
  The number and nature of adverse events (AEs) and series adverse events (SAEs) occurring during the study will be tracked and reported.
Time to Closure | 1-12 weeks
  Average number of grafts/weeks used to achieve wound closure
Follow-Up Closure | 2 weeks
  Number of wounds remaining closed during the 2-week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Desmond Bell, DPM, Study Chair — SygNola, LLC
Locations (5):
- United States (5):
  - MedCentris of Alexandria, Alexandria, Louisiana
  - MedCentris of Monroe, Monroe, Louisiana
  - MedCentris of Natchez, Natchez, Mississippi
  - MedCentris of Picayune, Picayune, Mississippi
  - Pace Foot and Ankle Center, Bryn Mawr, Pennsylvania

IPD SHARING:
Plan to Share IPD: No